CLINICAL TRIAL: NCT02318225
Title: Cervical Priming With Misoprostol Before Diagnostic Office Hysteroscopy in Patients With no Risk Factors for Experiencing Unacceptable Pain. A Randomized Double Blinded Placebo-controlled Study
Brief Title: Misoprostol Prior to Office Hysteroscopy in Patients With no Risk Factors for Experiencing Unacceptable Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Usama M Fouda, M.D, PhD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Miso/Placebo/hystero1
Record Dates: First submitted 2014-12-11; First posted 2014-12-17 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Misoprostol; Office hysteroscopy; Pain
MeSH Terms: conditions — Pain | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Active Comparator): Misoprostol (400µg) is administered vaginally 12 hours before office hysteroscopy
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Placebo is administered vaginally 12 hours before office hysteroscopy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — Misoprostol (400µg) will be administered vaginally 12 hours before office hysteroscopy. A rigid 2.9 mm hysteroscope with 30° forward oblique lens will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach as described by Betocchi and Selvaggi in 1997 . All the procedures will be diagnostic.
  Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used (zero indicates no pain and 10 indicates the worst possible experienced pain).
  Arms: Misoprostol
Drug: Placebo — Placebo will be administered vaginally 12 hours before office hysteroscopy. A rigid 2.9 mm hysteroscope with 30° forward oblique lens will be used in the procedure. The uterine cavity will be distended by warm saline at a pressure between 60-80 mmHg. All the procedures will be performed during the proliferative phase using the vaginoscopic approach as described by Betocchi and Selvaggi in 1997 . All the procedures will be diagnostic.
  Pain intensity will be assessed by visual analogue scale during the examination and 30 minutes after the procedure. A visual analogue scale ranging from 0 to 10 will be used (zero indicates no pain and 10 indicates the worst possible experienced pain).
  Arms: Placebo

SUMMARY:
The aim of this study is to assess whether vaginal misoprostol reduces pain during office hysteroscopy in parous patients with no risk factors for experiencing severe or unacceptable pain.

DETAILED DESCRIPTION:
Cervical ripening with misoprostol to minimize the pain experienced during office hysteroscopy has been proposed by several authors.

The use of misoprostol is usually associated with undesired side effects and therefore any beneficial effect of misoprostol on reducing pain should be weighed against its undesired side effects (nausea, vomiting, diarrhea, fever, shivering, pain) and coasts. Till now , no studies have yet determined whether misoprostol should be used routinely or for the subgroup of patients at higher risk for cervical stenosis.

The aim of this study is to assess whether vaginal misoprostol reduces pain during office hysteroscopy in parous patients with no risk factors for experiencing severe or unacceptable pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one vaginal delivery who have an indication for office hysteroscopy.

Exclusion Criteria:

* Nulliparous patients, menopausal patients and patients with cervical pathology, and previous history of caesarean section or cervical surgery

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | procedure

SECONDARY OUTCOMES:
Operative time | procedure

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D,PhD, Study Chair — Cairo University
Locations (1):
- Obstetrics and Gynecology Department,Cairo university, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Cicinelli E, Rossi AC, Marinaccio M, Matteo M, Saliani N, Tinelli R. Predictive factors for pain experienced at office fluid minihysteroscopy. J Minim Invasive Gynecol. 2007 Jul-Aug;14(4):485-8. doi: 10.1016/j.jmig.2007.03.008. PMID 17630168